CLINICAL TRIAL: NCT06403683
Title: Relationship Between Physical Activity Levels and Insomnia in Females With Primary Dysmenorrhea
Brief Title: Physical Activity Level and Insomnia
Status: Enrolling by invitation | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Adel Abdelaziz, Physiotherapy researcher, Cairo University
Other Study IDs: P.T.REC/012/004951
Record Dates: First submitted 2024-04-26; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Primary Dysmenorrhea
Keywords: Physical Activity Level; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Walk Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Females with primary dysmenorrhoea: 75 females complain from primary dysmenorrhoea according to WaLIDD score.
  Interventions: Diagnostic Test: WaLIDD score / Insomnia Severity Index (ISI) / International Physical Activity Questionnaire (Short-form) / Six-Minute Walk Test
- Females without primary dysmenorrhoea: 75 females don't complain from primary dysmenorrhoea according to WaLIDD score.
  Interventions: Diagnostic Test: WaLIDD score / Insomnia Severity Index (ISI) / International Physical Activity Questionnaire (Short-form) / Six-Minute Walk Test

INTERVENTIONS:
Diagnostic Test: WaLIDD score / Insomnia Severity Index (ISI) / International Physical Activity Questionnaire (Short-form) / Six-Minute Walk Test — Case control trial study

SUMMARY:
This study aims to investigate the relationship between physical activity levels and insomnia in females with primary dysmenorrhea.

DETAILED DESCRIPTION:
This study will be designed as a case-control study, conducted on 150 females recruited from El_Nassr hospital in Helwan, Cairo, Egypt and from social media. Patients will be divided into two equal groups: group A(75 patients complain from PD according to WaLIDD score)& group B(75 patients don't complain from PD according to WaLIDD score). All data and information of each female in this study, including name, age, address, weight, height, and menstrual history, will be recorded in a recording data sheet. WaLIDD score will be used to assess PD symptoms, Insomnia Severity Index will be used to assess insomnia, International Physical Activity Questionnaire (Short-form)& Six-Minute Walk Test will be used to assess physical activity levels. Inclusion criteria: 1)Patient ages will be ranged between 18-25 years old, 2)They do not receive any drugs, 3)Being a virgin. Participants will be excluded if they 1) Using hormonal contraception (such as oral contraceptives and injections), 2)Taking any medications, 3)History of chronic disease, 4)Having any psychiatric or gynecological problems (such as PCO, amenorrhea, women who suffered from menopause). The subject, who missed for any of assessment session, would be withdraw form the research.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ages will be ranged between 18-25 years old.
2. They do not receive any drugs.
3. Being a virgin .

Exclusion Criteria:

1. Using hormonal contraception (such as oral contraceptives and injections).
2. Taking any medications.
3. History of chronic disease.
4. Having any psychiatric or gynecological problems (such as PCO, amenorrhea, women who suffered from menopause).

Ages: 18 Years to 25 Years | Sex: Female
Age Groups: Adult
Study Population: This study will be conducted on 150 females recruited from El_ Nassr hospital in Helwan, Cairo, Egypt and from social media. Patients will be divided into two equal groups:
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Insomnia | Through study completion, an average of 6 months
  Record insomnia severity during menstruation
Physical activity level | Through study completion, an average of 6 months
  Record Physical activity level during menstruation

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Mohamed Kamel, PhD, Study Chair — Department of Woman's Health, Faculty of Physical Therapy, Cairo University, Giza, Egypt
Locations (1):
- Cairo University, Giza, Egypt